CLINICAL TRIAL: NCT05097794
Title: An Open-label, One-sequence, 3-period Study to Evaluate Drug-drug Interactions and Safety Between "BR1015-1" and "BR1015-2" in Healthy Volunteers.
Brief Title: A Clinical Trial to Evaluate Drug-drug Interactions and Safety Between "BR1015-1" and "BR1015-2" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BR-FMS-CT-118
Record Dates: First submitted 2021-10-17; First posted 2021-10-28 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Indapamide

STUDY DESIGN:
Intervention Model Description: One-sequence, 3-period study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence BR1015-1/BR1015-2/BR1015-1 + BR1015-2 (Experimental): A total of 32 subjects will be enrolled in one sequence group. The investigational products (IPs) will be administered according to the treatment groups(BR1015-1, BR1015-2, BR1015-1 + BR1015-2) assigned to one sequence group in Period 1, Period 2, and Period 3.
  * Period 1(BR1015-1): BR1015-1(Fimasartan 60mg) - 1 tablet QD, five-day repeated-dose
  * Period 2(BR1015-2): BR1015-2(Indapamide 1.5mg) - 1 tablet QD, five-day repeated-dose
  * Period 3(BR1015-1 + BR1015-2): BR1015-1 (Fimasartan 60mg) 1 tablet + BR1015-2 (Indapamide 1.5mg) 1 tablet QD, five-day repeated-dose
  * Washout period between Period 1 and Period 2: five days
  * Washout period between Period 2 and Period 3: two days
  Interventions: Drug: BR1015-1; Drug: BR1015-2; Drug: BR1015-1 + BR1015-2

INTERVENTIONS:
Drug: BR1015-1 — - Administration to the BR1015-1 group: 60 mg of BR1015-1 will be administered one tablet once a day, five-day repeated doses.
  Other Names: Fimasartan 60 mg
Drug: BR1015-2 — - Administration to the BR1015-2 group: 1.5 mg of BR1015-2 will be administered one tablet once a day, five-day repeated doses.
  Other Names: Indapamide 1.5 mg
Drug: BR1015-1 + BR1015-2 — - Co-administration to the BR1015-1+BR1015-2 group: 60 mg of BR1015-1 one tablet and 1.5 mg of BR1015-2 one tablet will be co-administered once a day, five-day repeated doses.
  Other Names: Fimasartan and Indapamide

SUMMARY:
The purpose of this study is to evaluate pharmacokinetic interactions (Drug-Drug interaction) and safety between "BR1015-1" and "BR1015-2" in healthy volunteers.

DETAILED DESCRIPTION:
*Study Objective: After repeated administration of BR1015-1 and BR1015-2 for healthy volunteers, the pharmacokinetic interactions and safety are evaluated.

*Investigational Product (and regimen)

1. BR1015-1: Administration of BR1015-1 60 mg once a day for 5 days
2. BR1015-2: Administration of BR1015-2 1.5 mg once a day for 5 days
3. BR1015-1+BR1015-2: Co-administration of BR1015-1 60 mg and BR1015-2 1.5 mg once a day for 5 days

ELIGIBILITY:
Inclusion Criteria:

* Subjects are given sufficient explanations about the trial objectives and contents as well as properties of investigational drugs before participating in the trial, and will voluntarily express their consent by signing an IRB-approved written consent to participate in the trial.
* Healthy adults aged 19 to 55 years at screening.
* The subject's weight is 50 kg or more for males, 45 kg or more for females, and body mass index (BMI) is 18.0 or more but 30.0 kg/m2 or less.

Exclusion Criteria:

* Those who have history of clinically significant diseases including hypersensitivity reaction, intolerability and anaphylaxis to major ingredients and other ingredients of investigational products.
* Those who have history of clinically significant diseases including allergy reaction to Yellow No. 5 (Sunset Yellow FCF).
* Those who have a history of clinically significant diseases related to liver, kidney, digestive system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, hemato-oncology system, cardiovascular system (including orthostatic hypotension), etc.
* Those who have medical history of gastrointestinal system diseases (for example: Crohn's disease, peptic ulcer disease, etc.) and operations that may influence the absorption of investigational drugs. (However, appendectomy, hernia operation, endoscopic polypectomy and hemorrhoids/anal fissure/anal fistula surgeries are excluded.)
* Those with abnormal findings from the screening tests (medical interview, vital signs, electrocardiography, physical checkup, blood test, urinalysis, etc.) are judged to have clinical significance.
* Those who are positive to HBsAg, HCV Ab, HIV Ab, VDRL tests at screening.
* Those with any of the following results at screening:
* AST or ALT > twice the upper limit of normal range
* T. bilirubin > twice the upper limit of normal range
* Estimated glomerular filtration rate (e-GFR) < 60 mL/min/1.73m2 (CKD-EPI method used)
* Na > 150 mEq/L or <130 mEq/L
* K > 5.5 mEq/L or <3.0 mEq/L
* Those with systolic blood pressure > 160 mmHg or < 110 mmHg, or diastolic blood pressure > 100 mmHg or < 70 mmHg from vital signs at screening.
* Others who are judged to be ineligible to participate in the trial by the investigator.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
[Part A] Cmax,ss of BR1015-1 | 0~24 hour after administration at Day 5.
  Pharmacokinetic variables - Maximum (peak) plasma concentration of BR1015-1 at steady state (Cmax,ss).
[Part B] Cmax,ss of BR1015-2 | 0~24 hour after administration at Day 5.
  Pharmacokinetic variables - Maximum (peak) plasma concentration of BR1015-2 at steady state (Cmax,ss).
[Part A] AUCtau of BR1015-1 | 0~24 hour after administration at Day 5.
  Pharmacokinetic variables - Area under the plasma drug concentration-time curve to the end of the dosing period in multiple dosing of BR1015-1 at steady state. (AUCtau,ss)
[Part B] AUCtau of BR1015-2 | 0~24 hour after administration at Day 5.
  Pharmacokinetic variables - Area under the plasma drug concentration-time curve to the end of the dosing period in multiple dosing of BR1015-2 at steady state. (AUCtau,ss)

SECONDARY OUTCOMES:
[Part A] AUClast of BR1015-1 | 0~48 hour after administration
  Area under the plasma drug concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration (AUClast) of BR1015-1
[Part B] AUClast of BR1015-2 | 0~48 hour after administration
  Area under the plasma drug concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration (AUClast) of BR1015-2
[Part A] AUCinf of BR1015-1 | 0~48 hour after administration
  Area under the plasma drug concentration-time curve over the time interval from 0 extrapolated to infinity of BR1015-1
[Part B] AUCinf of BR1015-2 | 0~48 hour after administration
  Area under the plasma drug concentration-time curve over the time interval from 0 extrapolated to infinity of BR1015-2
[Part A] Tmax of BR1015-1 | 0~24 hour after administration
  Time to reach maximum (peak) plasma concentration following drug administration at steady state (Tmax,ss)
[Part B] Tmax of BR1015-2 | 0~24 hour after administration
  Time to reach maximum (peak) plasma concentration following drug administration at steady state (Tmax,ss)
[Part A] t1/2 of BR1015-1 | 0~48 hour after administration
  Terminal half-life of BR1015-1
[Part B] t1/2 of BR1015-2 | 0~48 hour after administration
  Terminal half-life of BR1015-2

CONTACTS AND LOCATIONS:
Overall Officials: An-Hye Kim, M.D. Ph.D, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Gyeonggi-do, Seongnam-si, South Korea